CLINICAL TRIAL: NCT03874429
Title: Comparison of the Performance and Safety of T2259 Versus Vismed Multi in Dry Eye Patients With Superficial Keratitis.
Brief Title: Efficacy of T2259 in DED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2259-001
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Masking Description: investigator-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2259 (Experimental): 1 drop in each eye 2 to 4 times daily
  Interventions: Device: T2259
- Vismed Multi (Active Comparator): 1 drop in each eye 2 to 4 times daily
  Interventions: Device: Vismed multi

INTERVENTIONS:
Device: T2259 — Sodium Hyaluronate and Trehalose
  Other Names: Sodium Hyaluronate and Trehalose
  Arms: T2259
Device: Vismed multi — HA
  Other Names: Sodium Hyaluronate
  Arms: Vismed Multi

SUMMARY:
The purpose of this study is to compare the performance and safety of T2259 versus Vismed Multi in dry eye patients with superficial keratitis.

ELIGIBILITY:
Main inclusion Criteria:

* Signed and dated informed consent
* Male or female aged from ≥ 18 years old
* Known Dry Eye Syndrome requiring artificial tears within the last 3 months prior to study selection

Main exclusion Criteria:

* Far best-corrected visual acuity≤2/10
* Severe Blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.N.O des XV-XX, Paris, France

RESULTS

PARTICIPANT FLOW:
Groups:
- T2259; Vismed Multi: 1 drop in each eye 2 to 4 times daily 3 months treatment period lasted from randomisation visit (Day 1 ; Visit #2) to the final visit (Day 84 (7 days) ; Visit #5)
Period: Overall Study
Arm/Group | T2259 | Vismed Multi
Started | 50 | 51
Completed | 44 | 46
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Covid-19 pandemic | 4 | 2

BASELINE CHARACTERISTICS:
Population: FAS population
Groups:
- T2259: 1 drop in each eye 2 to 4 times daily
  T2259
- Vismed Multi: 1 drop in each eye 2 to 4 times daily
  Vismed multi
- Total: Total of all reporting groups
Arm/Group | T2259 | Vismed Multi | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 41 | 65
  >=65 years | 25 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 62.4 (13.7) | 55.5 (13.1) | 59 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 87
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 11 | 8 | 19
  Spain | 12 | 10 | 22
  Poland | 4 | 6 | 10
  Slovakia | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Surface Ocular Staining With Fluorescein (With Oxford Scale - Ranges : 0-15)
Description: Change from baseline in the worse eye at Day 35 in Global Ocular staining (decrease of oxford score = better outcome)
Time Frame: Baseline and Day 35
Population: PP population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T2259 | Vismed Multi
Number analyzed (Participants) | 42 | 42
score on a scale | -1.45 (1.88) | -1.79 (1.68)
Statistical Analysis 1: Comparison: T2259 vs Vismed Multi; To assess the non inferiority of T2259 compared to Vismed Multi, two-sided 95% confidence interval from ANCOVA model was computed of the difference of T2259 minus Vismed Multi. The model was adjusted for the main effects of investigation product and baseline score; Test type: Non-Inferiority — Non- inferiority was demonstrated if the upper bound of the 95% CI was no higher than 2 points for the the difference of T2259 minus Vismed Multi; ANCOVA; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.42 to 1.05], Standard Error of Mean 0.37

ADVERSE EVENTS:
Time Frame: 15 weeks from D-10 to D84 (±7 days)
Arm/Group | T2259 | Vismed Multi
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/51
Other Adverse Events (participants affected / at risk) | 4/50 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T2259 (N=50) | Vismed Multi (N=51)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T2259 (N=50) | Vismed Multi (N=51)
Headache (Nervous system disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03874429/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03874429/SAP_001.pdf